CLINICAL TRIAL: NCT04177108
Title: A Phase III, Double-blind, Placebo-controlled, Randomized Study of Ipatasertib in Combination With Atezolizumab and Paclitaxel as a Treatment for Patients With Locally Advanced Unresectable or Metastatic Triple-Negative Breast Cancer
Brief Title: A Study of Ipatasertib in Combination With Atezolizumab and Paclitaxel as a Treatment for Participants With Locally Advanced or Metastatic Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CO41101; 2019-000810-12 (EudraCT Number)
Record Dates: First submitted 2019-11-07; First posted 2019-11-26 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Triple-Negative Breast Cancer
Keywords: Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Skin Diseases; Paclitaxel; Atezolizumab; Ipatasertib; Antibodies, Monoclonal; Antineoplastic Agents, Phytogenic; Antineoplastic Agents; Tubulin Modulators; Antimitotic Agents; Mitosis Modulators
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Skin Diseases | interventions — atezolizumab; ipatasertib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel (Experimental): TNBC participants with programmed death-ligand 1 (PD-L1) non-positive received a combination of paclitaxel, 80 milligrams per meter square (mg/m^2), intravenous (IV) infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, 400 mg, orally (PO), once daily (QD), from Day 1 to Day 21 of each 28-day cycle and atezolizumab, 840 mg, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
  Interventions: Drug: Atezolizumab; Drug: Ipatasertib; Drug: Paclitaxel
- Cohort 1 Arm B: Ipatasertib + Placebo + Paclitaxel (Experimental): TNBC participants with PD-L1 non-positive received a combination of paclitaxel, 80 mg/m^2, IV infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, 400 mg, PO, QD, from Day 1 to Day 21 of each 28-day cycle and atezolizumab-matching placebo, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
  Interventions: Drug: Ipatasertib; Drug: Paclitaxel; Drug: Placebo for Atezolizumab
- Cohort 1 Arm C: Placebo + Placebo + Paclitaxel (Experimental): TNBC participants with PD-L1 non-positive received a combination of paclitaxel, 80 mg/m^2, IV infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib-matching placebo, PO, QD, from Day 1 to Day 21 of each 28-day cycle and atezolizumab-matching placebo, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
  Interventions: Drug: Paclitaxel; Drug: Placebo for Atezolizumab; Drug: Placebo for Ipatasertib
- Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxel (Experimental): TNBC participants with PD-L1 positive received a combination of paclitaxel, 80 mg/m^2, IV infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, 400 mg, PO, QD, from Day 1 to Day 21 of each 28-day cycle and atezolizumab, 840 mg, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
  Interventions: Drug: Atezolizumab; Drug: Ipatasertib; Drug: Paclitaxel
- Cohort 2 Arm B: Placebo+ Atezolizumab + Paclitaxel (Experimental): TNBC participants with PD-L1 positive received a combination of paclitaxel, 80 mg/m^2, IV infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib-matching placebo, PO, QD, from Day 1 to Day 21 of each 28-day cycle and atezolizumab, 840 mg, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
  Interventions: Drug: Atezolizumab; Drug: Paclitaxel; Drug: Placebo for Ipatasertib

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab was administered as per the dosage regimen mentioned in arm descriptions.
  Arms: Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel; Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxel; Cohort 2 Arm B: Placebo+ Atezolizumab + Paclitaxel
Drug: Ipatasertib — Ipatasertib was administered as per the dosage regimen mentioned in arm descriptions.
  Arms: Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel; Cohort 1 Arm B: Ipatasertib + Placebo + Paclitaxel; Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxel
Drug: Paclitaxel — Paclitaxel was administered as per the dosage regimen mentioned in arm descriptions.
Drug: Placebo for Atezolizumab — Placebo was administered as per the dosage regimen mentioned in arm descriptions.
  Arms: Cohort 1 Arm B: Ipatasertib + Placebo + Paclitaxel; Cohort 1 Arm C: Placebo + Placebo + Paclitaxel
Drug: Placebo for Ipatasertib — Placebo was administered as per the dosage regimen mentioned in arm descriptions.
  Arms: Cohort 1 Arm C: Placebo + Placebo + Paclitaxel; Cohort 2 Arm B: Placebo+ Atezolizumab + Paclitaxel

SUMMARY:
This study evaluated the efficacy and safety of ipatasertib in combination with atezolizumab and paclitaxel in locally advanced or metastatic Triple-Negative Breast Cancer (TNBC) previously untreated in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness and ability to complete all study-related assessments, including Participant-Reported Outcome (PRO) assessments, in the investigator's judgement.
2. Adequate hematologic and organ function within 14 days before the first study treatment on Day 1 of Cycle 1.
3. Life expectancy of at least 6 months.
4. Measurable disease according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v 1.1).
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs.
7. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating sperm.
8. Appropriate candidate for paclitaxel monotherapy if tumor programmed death-ligand 1 (PD-L1) status is unknown or non-positive; appropriate candidate for paclitaxel and atezolizumab if tumor PD-L1 status is positive.
9. Histologically documented triple-negative adenocarcinoma of the breast that is locally advanced or metastatic and is not amenable to resection with curative intent.

Exclusion Criteria:

1. Inability to comply with study and follow-up procedures.
2. History of malabsorption syndrome or other condition that would interfere with enteral absorption or results in the inability or unwillingness to swallow pills.
3. Severe infection within 4 weeks prior to initiation of study treatment (including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia) as well as those who have received treatment with therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to initiation of study treatment.
4. Known human immunodeficiency virus (HIV) infection (there must be a negative HIV test at screening).
5. Known clinically significant history of liver disease consistent with Child-Pugh Class B or C.
6. Current treatment with anti-viral therapy for hepatitis B virus (HBV).
7. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of Cycle 1 or anticipation of need for a major surgical procedure during the study.
8. Pregnancy or breastfeeding, or intention to become pregnant during the study or within 28 days after the final dose of ipatasertib or (/) placebo, 5 months after the final dose of atezolizumab/placebo, and 6 months after the final dose of paclitaxel whichever occurs later.
9. New York Heart Association Class II, III, or IV heart failure, left ventricular ejection fraction less than (<) 50 percent (%), or active ventricular arrhythmia requiring medication.
10. Current unstable angina or history of myocardial infarction within 6 months prior to Day 1 of Cycle 1.
11. Congenital long QT syndrome or screening QT interval corrected through use Fridericia's formula (QTcF) greater than (>) 480 milliseconds (ms).
12. Current treatment with medications used at doses known to cause clinically relevant prolongation of QT/QTc interval.
13. History or presence of an abnormal ECG that is clinically significant in the investigator's opinion (including complete left bundle branch block, second- or third-degree heart block, or evidence of prior myocardial infarction).
14. Requirement for chronic corticosteroid therapy of > 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids or immunosuppressant agents for a chronic disease.
15. Treatment with approved or investigational cancer therapy within 14 days prior to Day 1 of Cycle 1.
16. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the participant at high risk from treatment complications.
17. History of or known presence of spinal cord metastases, as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening or prior radiographic assessments.
18. Known central nervous system (CNS) disease, except for treated asymptomatic CNS metastases.
19. Known germline breast cancer gene (BRCA)1/2 deleterious mutation, unless the participant is not an appropriate candidate for a poly adenosine diphosphate ribose polymerase (PARP)-inhibitor.
20. Any previous systemic therapy for inoperable locally advanced or metastatic triple-negative adenocarcinoma of the breast.
21. Unresolved, clinically significant toxicity from prior therapy, except for alopecia and Grade 1 peripheral neuropathy.
22. Participants who have received palliative radiotherapy to peripheral sites (e.g., bone metastases) for pain control and whose last treatment was completed 14 days prior to Day 1 of Cycle 1 may be enrolled in the study if they have recovered from all acute, reversible effects (e.g., to Grade 1 or resolved by enrolment).
23. Uncontrolled pleural effusion, pericardial effusion or ascites.
24. Uncontrolled tumor-related pain.
25. Malignancies other than breast cancer within 5 years prior to Day 1 of Cycle 1, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer.
26. Known hypersensitivity or contraindication to any component of the study treatments, including the paclitaxel excipient, macrogolglycerol ricinoleate.
27. Grade greater than or equal to (≥) 2 peripheral neuropathy.
28. History of Type I or Type II diabetes mellitus requiring insulin.
29. Grade ≥ 2 uncontrolled or untreated hypercholesterolemia or hypertriglyceridemia.
30. History of or active inflammatory bowel disease (e.g., Crohn disease and ulcerative colitis) or active bowel inflammation (e.g., diverticulitis).
31. Lung disease: pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, Aspergillosis, active tuberculosis, or history of opportunistic infections (pneumocystis pneumonia or cytomegalovirus pneumonia).
32. Treatment with strong Cytochrome P450 (CYP)3A inhibitors or strong CYP3A inducers within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug.
33. Prior treatment with an Protein kinase B (Akt) inhibitor.
34. Active or history of autoimmune disease or immune deficiency.
35. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
36. Prior allogeneic stem cell or solid organ transplantation.
37. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during treatment with atezolizumab or within 5 months after the final dose of atezolizumab.
38. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
39. Known hypersensitivity to Chinese hamster ovary cell products or recombinant human antibodies.
40. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin-2) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment.
41. Treatment with systemic immunosuppressive medication (including, but not limited to corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (182):
- United States (31):
  - USA Mitchell Cancer Institute, Mobile, Alabama
  - Highlands Oncology Group, Springdale, Arkansas
  - UCLA, Los Angeles, California
  - Kaiser Permanente-SCPMG; Oncology Research, San Diego, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente - Franklin, Denver, Colorado
  - Stamford Hospital; BCC, MOHR, Stamford, Connecticut
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Healthcare System - Memorial Regional Hospital, Hollywood, Florida
  - Memorial Cancer Institute at Memorial West, Pembroke Pines, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Nancy N. and J.C. Lewis Cancer & Research Pavillion -St. Josephs / Candler Health System-CCD PRIME, Savannah, Georgia
  - Rush University, Chicago, Illinois
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Ochsner Health System, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Medstar Franklin Square Medical Center, Baltimore, Maryland
  - St. Joseph Mercy Hospital; Cancer Care Center., Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - CHI Health Saint Francis; Oncology, Grand Island, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack Univ Med Ctr, Hackensack, New Jersey
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Kaiser Permanente - Portland, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Charleston Oncology, P .A, Charleston, South Carolina
  - Greenville Health System; Cancer Center, Greenville, South Carolina
  - The West Clinic; West Cancer Center, Germantown, Tennessee
  - Vanderbilt Univ Medical Ctr, Nashville, Tennessee
- Argentina (6):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Inst. Angel Roffo; Haematology, Buenos Aires
  - Hospital Britanico, Ciudad Autonoma Bs As
  - Instituto Medico Rio Cuarto, Córdoba
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Fundacion Scherbovsky, Mendoza
- Australia (10):
  - Macquarie University Hospital, Macquarie Park, New South Wales
  - Mid North Coast Cancer Institute, Port Macquarie, New South Wales
  - Royal North Shore Hospital; Department of Medical Oncology, St Leonards, New South Wales
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Monash Health Monash Medical Centre, Clayton, Victoria
  - Peter MacCallum Cancer Centre; Medical Oncology, Melbourne, Victoria
  - Sunshine Hospital; Oncology Research, St Albans, Victoria
  - St John of God Hospital; Bendat Cancer Centre, Subiaco, Western Australia
- Austria (4):
  - Tiroler Landeskrankenanstalten Ges.M.B.H.; Abt. Für Gynäkologie, Innsbruck
  - Ordensklinikum Linz Barmherzige Schwestern; Interne 1 - Hämato-Onkologie, Linz
  - Uniklinikum Salzburg, LKH; Univ.Klinik f. Innere Medizin III der PMU, Salzburg
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I, Vienna
- Belgium (2):
  - AZ Maria Middelares, Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
- Brazil (4):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
  - Núcleo de Pesquisa São Camilo; ONCOLOGIA CLINICA / QUIMIOTERAPIA, São Paulo, São Paulo
- MHAT Nadezhda, Sofia, Bulgaria
- Canada (8):
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - Fraser Valley Centre British Columbia Cancer Agency, Surrey, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Royal Victoria Hospital, Barrie, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Jewish General Hospital; Research Unit, Montreal, Quebec
  - McGill University; Glen Site; Oncology, Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
- Colombia (2):
  - Clinica del Country, Bogotá
  - Oncólogos de Occidente, Pereira
- Clinica CIMCA, San José, Costa Rica
- Czechia (2):
  - Masaryk?v onkologický ústav; Klinika komplexní onkologické pé?e, Brno
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
- Denmark (2):
  - Herlev Hospital; Afdeling for Kræftbehandling, Herlev
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
- Finland (3):
  - Docrates Cance Center, Helsinki
  - KYS Sadesairaala; Syopatautien poliklinikka, Kuopio
  - VAASAN KESKUSSAIRAALA; Onkologian poliklinikka, Vaasa
- Centre Eugene Marquis; Service d'oncologie, Rennes, France
- Greece (2):
  - Agioi Anargyroi Cancer Hospital; 2Nd Oncology Dept., Kifissia
  - Euromedical General Clinic of Thessaloniki; Oncology Department, Thessaloniki
- Hong Kong (3):
  - Queen Mary Hospital; Dept of Medicine, Hong Kong
  - Tuen Mun Hospital; Clinical Onc, Hong Kong
  - Prince of Wales Hospital; Department of Clinical Onocology, Shatin
- Sahyadri Super Specialty Hospital Hadapsar, Pune, Maharashtra, India
- Shaare Zedek Medical Center, Jerusalem, Israel
- Italy (8):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - ASU FC S. M. DELLA MISERICORDIA; Oncologia, Udine, Friuli Venezia Giulia
  - ASST DEGLI SPEDALI CIVILI DI BRESCIA; Oncologia Medica, Brescia, Lombardy
  - ASST DI LECCO; Oncologia Medica, Lecco, Lombardy
  - IRCCS Istituto Clinico Humanitas; Oncologia, Rozzano (MI), Lombardy
  - Ospedale Civile; Unita Operativa Di Oncologia Medica, Livorno, Tuscany
  - IOV - Istituto Oncologico Veneto - IRCCS; Oncologia Medica II, Padua, Veneto
- Japan (8):
  - Aichi Cancer Center Hospital, Aichi
  - Fukushima Medical University Hospital, Fukushima
  - Gunma Prefectural Cancer Center, Gunma
  - Hiroshima University Hospital, Hiroshima
  - Kanagawa Cancer Center, Kanagawa
  - Kumamoto Shinto General Hospital, Kumamoto
  - Okayama University Hospital, Okayama
  - Osaka International Cancer Institute, Osaka
- Mexico (3):
  - Investigacion Oncofarmaceutica, La Paz, Baja California Sur
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Christus Muguerza Clinica Vidriera, Monterrey, Nuevo León
- New Zealand (3):
  - Auckland City Hospital, Cancer and Blood Research, Auckland
  - Tauranga Hospital, Clinical Trials Unit; BOP Clinical School, Tauranga
  - Wellington Regional Hospital; Clinical Trials Unit, Wellington
- Peru (8):
  - Centro Medico Monte Carmelo, Arequipa
  - Instituto Regional de Enfermedades Neoplasicas, Arequipa
  - Unidad de Investigación Oncologica; Hospital Nacional Daniel Alcides Carrion, Lima
  - Clínica San Gabriel; Unidad de Investigación Oncológica de la Clínica San Gabriel, Lima
  - Hospital Arzobispo Loayza, Lima
  - Oncosalud Sac; Oncología, Lima
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Clinica Ricardo Palma, San Isidro
- Poland (5):
  - Instyt. Centrum Zdrowia Matki Polki; Klinika Chirurgii Onk. Chorób Piersi z Podod. Onko Klinicznej, ?ód?
  - Narodowy Inst.Onkol.im.Sklodowskiej-Curie Panstw.Inst.Bad Gliwice; Centr.Diagn.i Lecz.Chor.Piersi, Gliwice
  - Szpital Uniwersytecki w Krakowie, Oddzia? Kliniczny Kliniki Onkologii, Krakow
  - Wielkopolskie Centrum Onkologii, Poznan
  - Narodowy Instytut Onkologii im. M.Sklodowskiej-Curie; Klinika Nowotworow Piersi i Chirurgii Rekonstr, Warsaw
- Portugal (5):
  - Hospital da Luz; Departamento de Oncologia Medica, Lisbon
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - Hospital Beatriz Angelo; Departamento de Oncologia, Loures
  - Centro Hospitalar do Porto ? Hospital de Santo António; Oncologia, Porto
  - IPO do Porto; Servico de Oncologia Medica, Porto
- Oncology Center Sf. Nectarie, Craiova, Romania
- Russia (9):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arhangelsk
  - University ?linic of headaches, Moscow, Moscow Oblast
  - P.A. Gertsen Cancer Research Inst. ; Chemotherapy Dept, Moscow, Moscow Oblast
  - SBIH "Moscow Clinical Scientific and Practical Center named after A.S. Loginov of DHM", Moskva, Moscow Oblast
  - Fed State Budgetary Inst "N.N. Blokhin Med Center of Oncology" MHRF, Moskva, Moscow Oblast
  - FSAI Treatment and rehabilitation Centre Ministry of Health; Clinical research and chemotherapy., Moskva, Moscow Oblast
  - S-Pb clinical scientific practical center of specialized kinds of medical care (oncological), Saint Petersburg, Sankt-Peterburg
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan', Tatarstan Republic
  - Limited Liability Company "RC Medical", Novosibirsk
- National Cancer Centre; Medical Oncology, Singapore, Singapore
- South Africa (5):
  - National Hospital; Oncotherapy Dept, Bloemfontein
  - Cancercare, George
  - Wits Clinical Research, Johannesberg
  - Cancercare, Port Elizabeth
  - Wilgers Oncology Centre, Pretoria
- South Korea (6):
  - Kyungpook National University Medical Center, Daegu
  - National Cancer Center, Goyang-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
- Spain (11):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Hospital Provincial de Castellon; Servicio de Oncologia, Castellon, Castellon
  - Complejo Hospitalario Universitario A Coruña (CHUAC); Servicio de Oncologia, A Coruña, LA Coruña
  - Hospital Universitario Puerta de Hierro; Servicio de Oncologia, Majadahonda, Madrid
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal; Servicio de Oncología, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Clínico Universitario de Valencia; Servicio de Oncología, Valencia
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Universitätsspital Zürich Gynäkologische Klinik; Klinik für Gynäkologie, Zurich
- Taiwan (4):
  - China Medical University Hospital; Surgery, Taichung
  - VETERANS GENERAL HOSPITAL; Department of General Surgery, Taipei
  - National Taiwan Uni Hospital; General Surgery, Taipei
  - Chang Gung Memorial Hosipital at Linkou, Taoyuan
- Thailand (6):
  - Chulalongkorn Hospital; Medical Oncology, Bangkok
  - Rajavithi Hospital; Division of Medical Oncology, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital; Department of Surgery/Head Neck and Breast Unit; Clinical Trial, Chiang Mai
  - Khonkaen Hospital, Khonkaen
  - Songklanagarind Hospital; Department of Oncology, Songkhla
- Turkey (Türkiye) (3):
  - Memorial Ankara Hastanesi, Ankara
  - Medipol University Medical Faculty; Oncology Department, Istanbul
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sihhiye/Ankara
- Ukraine (7):
  - SI Institute of general&urgent surgery n/a Zaytseva V.T NAMSU; Purulent Surgery department, Kharkiv, Kharkiv Governorate
  - Regional Oncology Center; Department of Mammology, Chernihiv
  - Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipropetrovsk
  - ME Kryviy Rih Oncology Dispensary of Dnipropetrovs?k Regional Council; Chemotherapy Department, Kryvyi Rih
  - MI Kyiv Regional Council Kyiv Regional Oncological Dispensary; Department of Mammology, Kyiv
  - Municipal Institution Odesa Regional Clinical Hospital, Odesa
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
- United Kingdom (3):
  - BEATSON WEST OF SCOTLAND CANCER CENTRE; Clinical Research Unit ? Level 1, Glasgow
  - The Royal Marsden Hospital, Fulham, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 215 investigative centers from 25 November 2019 to 28 February 2023.
Pre-assignment Details: A total of 242 participants with Advanced triple-negative breast cancer (TNBC) were enrolled, of which 127 participants were randomized to cohort 1 {programmed death-ligand 1 (PD-L1) Non-positive} and 115 participants to cohort 2 (PD-L1 positive).
Groups:
- Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel: TNBC participants with PD-L1 non-positive received a combination of paclitaxel, 80 milligrams per meter square (mg/m^2), intravenous (IV) infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, 400 mg, orally (PO), once daily (QD), from Day 1 to Day 21 of each 28-day cycle and atezolizumab, 840 mg, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
- Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel: TNBC participants with PD-L1 non-positive received a combination of paclitaxel, 80 mg/m^2, IV infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, 400 mg, PO, QD, from Day 1 to Day 21 of each 28-day cycle and atezolizumab-matching placebo, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
- Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel: TNBC participants with PD-L1 non-positive received a combination of paclitaxel, 80 mg/m^2, IV infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib-matching placebo, PO, QD, from Day 1 to Day 21 of each 28-day cycle and atezolizumab-matching placebo, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
- Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel: TNBC participants with PD-L1 positive received a combination of paclitaxel, 80 mg/m^2, IV infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib-matching placebo, PO, QD, from Day 1 to Day 21 of each 28-day cycle and atezolizumab, 840 mg, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
Period: Overall Study
Arm/Group | Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel | Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel | Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel
Started | 43 | 43 | 41 | 58 | 57
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 43 | 43 | 41 | 58 | 57
Not completed — Withdrawal by Subject | 4 | 8 | 9 | 11 | 13
Not completed — Physician Decision | 23 | 15 | 18 | 29 | 23
Not completed — Reason Not Specified | 0 | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1
Not completed — Death | 16 | 19 | 13 | 17 | 18

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants randomized in this study.
Groups:
- Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel: TNBC participants with PD-L1 non-positive received a combination of paclitaxel, 80 mg/m^2, IV infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, 400 mg, PO, QD, from Day 1 to Day 21 of each 28-day cycle and atezolizumab, 840 mg, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel | Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel | Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel | Total
Number analyzed (Participants) | 43 | 43 | 41 | 58 | 57 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.7) | 50.8 (11.6) | 53.5 (10.7) | 53.7 (12.1) | 51.1 (11.7) | 52.9 (11.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 43 | 43 | 41 | 58 | 57 | 242
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 6 | 15 | 14 | 52
  Not Hispanic or Latino | 32 | 32 | 35 | 41 | 43 | 183
  Unknown or Not Reported | 3 | 2 | 0 | 2 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 1 | 5 | 6 | 20
  Asian | 10 | 7 | 9 | 19 | 16 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 2 | 2 | 8
  White | 26 | 29 | 29 | 29 | 32 | 145
  More than one race | 0 | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 2 | 1 | 3 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS was defined as the time from randomization to the first occurrence of disease progression as determined locally by RECIST or death from any cause during treatment, whichever occurs first.
Time Frame: From Randomization to disease progression, study completion, or death (up to 39 months)
Population: ITT population included all participants randomized in this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel | Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel | Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel
Number analyzed (Participants) | 43 | 43 | 41 | 58 | 57
months | 7.1 [5.1 to 9.3] | 5.6 [3.7 to 8.2] | 3.7 [3.6 to 5.4] | 5.6 [5.4 to 9.2] | 5.7 [4.0 to 9.1]
Statistical Analysis 1: Comparison: Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel vs Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel; Test type: Superiority; p = 0.0098, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI [0.28 to 0.85]
Statistical Analysis 2: Comparison: Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel vs Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel; Test type: Superiority; p = 0.2396, Log Rank; Hazard Ratio (HR) = 0.72, 95% CI [0.42 to 1.25]
Statistical Analysis 3: Comparison: Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxel vs Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel; Test type: Superiority; p = 0.9809, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI [0.63 to 1.58]

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the time of death from any cause on study.
Time Frame: From randomization up to study completion or death (Up to 39 months)
Population: ITT population included all participants randomized in this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel | Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel | Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel
Number analyzed (Participants) | 43 | 43 | 41 | 58 | 57
months | 15.7 [12.5 to NA] — Upper limit of 95% confidence interval (CI) could not be calculated due to insufficient number of participants with events. | 15.3 [15.3 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 16.6 [9.6 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | NA [14.1 to NA] — Median and upper limit of 95% CI could not be calculated due to insufficient number of participants with events. | 17.2 [13.4 to NA] — Upper limit of 95% CI could not be calculated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel vs Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel; Test type: Superiority; p = 0.6805, Log Rank; Hazard Ratio (HR) = 1.17, 95% CI [0.55 to 2.51]
Statistical Analysis 2: Comparison: Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel vs Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel; Test type: Superiority; p = 0.6314, Log Rank; Hazard Ratio (HR) = 1.21, 95% CI [0.55 to 2.64]
Statistical Analysis 3: Comparison: Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxel vs Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel; Test type: Superiority; p = 0.9164, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI [0.52 to 2.06]

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Up to 39 months
Population: Safety-evaluable population included all randomized participants who took at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel | Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel | Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel
Number analyzed (Participants) | 43 | 43 | 41 | 58 | 57
Participants | 42 | 43 | 40 | 58 | 56

ADVERSE EVENTS:
Time Frame: Up to 39 months
Description: Safety-evaluable population included all randomized participants who took at least one dose of the study treatment.
Groups:
- Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxe: TNBC participants with PD-L1 positive received a combination of paclitaxel, 80 mg/m^2, IV infusion on Days 1, 8, and 15 of each 28-day cycle and ipatasertib, 400 mg, PO, QD, from Day 1 to Day 21 of each 28-day cycle and atezolizumab, 840 mg, IV infusion on Day 1 and 15 of each 28-day cycle until loss of clinical benefit, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
Arm/Group | Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel | Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel | Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel | Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxe | Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 16/43 | 19/43 | 13/41 | 18/58 | 18/57
Serious Adverse Events (participants affected / at risk) | 14/43 | 7/43 | 7/41 | 16/58 | 9/57
Other Adverse Events (participants affected / at risk) | 42/43 | 42/43 | 40/41 | 56/58 | 55/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel (N=43) | Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel (N=43) | Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel (N=41) | Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxe (N=58) | Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel (N=57)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vocal cord atrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 Arm A: Ipatasertib + Atezolizumab + Paclitaxel (N=43) | Cohort 1 Arm B: Ipatasertib + Atezolizumab Matching Placebo + Paclitaxel (N=43) | Cohort 1 Arm C: Ipatasertib Matching Placebo + Atezolizumab Matching Placebo + Paclitaxel (N=41) | Cohort 2 Arm A: Ipatasertib + Atezolizumab + Paclitaxe (N=58) | Cohort 2 Arm B: Ipatasertib Matching Placebo+ Atezolizumab + Paclitaxel (N=57)
Anaemia (Blood and lymphatic system disorders) | 15 (22) | 7 (18) | 6 (10) | 22 (36) | 12 (17)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 2 (2) | 2 (6) | 8 (13) | 4 (7)
Neutropenia (Blood and lymphatic system disorders) | 15 (21) | 5 (21) | 8 (26) | 11 (36) | 9 (19)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2) | 0 (0) | 6 (7) | 6 (7)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (4) | 4 (5) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (7) | 0 (0) | 2 (2) | 5 (7) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7) | 12 (16) | 26 (29) | 16 (22) | 24 (33)
Diarrhoea (Gastrointestinal disorders) | 32 (66) | 30 (71) | 15 (22) | 37 (81) | 16 (28)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 3 (3) | 2 (2) | 6 (8) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 17 (21) | 14 (16) | 9 (10) | 22 (36) | 13 (16)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 6 (7) | 2 (3) | 7 (8) | 3 (4)
Vomiting (Gastrointestinal disorders) | 7 (16) | 10 (14) | 0 (0) | 8 (10) | 8 (9)
Asthenia (General disorders) | 9 (10) | 6 (8) | 7 (9) | 13 (24) | 5 (5)
Fatigue (General disorders) | 8 (12) | 10 (12) | 5 (8) | 14 (15) | 11 (11)
Mucosal inflammation (General disorders) | 6 (7) | 3 (3) | 0 (0) | 4 (5) | 6 (7)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 4 (6) | 4 (5) | 1 (3)
Pain (General disorders) | 0 (0) | 1 (1) | 3 (4) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 6 (6) | 3 (5) | 1 (2) | 7 (10) | 7 (8)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (4) | 2 (8) | 3 (3) | 2 (3)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 4 (5) | 1 (1) | 3 (8) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (5) | 1 (2) | 2 (2) | 8 (11) | 5 (7)
Alanine aminotransferase increased (Investigations) | 11 (15) | 11 (12) | 12 (15) | 12 (19) | 11 (18)
Aspartate aminotransferase increased (Investigations) | 7 (9) | 10 (14) | 10 (18) | 11 (16) | 10 (18)
Blood alkaline phosphatase increased (Investigations) | 5 (7) | 6 (9) | 1 (1) | 6 (9) | 1 (1)
Blood creatinine increased (Investigations) | 5 (7) | 2 (2) | 0 (0) | 5 (8) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 6 (14) | 1 (1) | 3 (7) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 4 (5) | 2 (4) | 0 (0) | 6 (7) | 1 (1)
Lipase increased (Investigations) | 1 (4) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (16) | 1 (9) | 0 (0) | 3 (10) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (12) | 9 (14) | 5 (7) | 9 (20) | 6 (16)
Weight decreased (Investigations) | 4 (4) | 0 (0) | 1 (2) | 3 (3) | 1 (1)
White blood cell count decreased (Investigations) | 5 (13) | 6 (14) | 1 (2) | 4 (11) | 2 (10)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7) | 6 (6) | 6 (7) | 16 (20) | 7 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (12) | 4 (9) | 2 (2) | 12 (18) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 3 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (11) | 0 (0) | 5 (5) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 0 (0) | 1 (1) | 6 (8) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 4 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5) | 3 (3) | 7 (8) | 4 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5) | 2 (2) | 5 (7) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 2 (2) | 5 (5) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 8 (9) | 9 (26) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4) | 4 (4) | 2 (11) | 5 (5) | 4 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 7 (8) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 6 (6) | 3 (3) | 11 (15) | 12 (14)
Neuropathy peripheral (Nervous system disorders) | 15 (19) | 8 (9) | 10 (11) | 8 (8) | 8 (9)
Paraesthesia (Nervous system disorders) | 5 (6) | 3 (3) | 3 (3) | 4 (5) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 6 (7) | 5 (6) | 11 (11) | 9 (10)
Polyneuropathy (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (6) | 3 (3) | 6 (6) | 4 (4)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 0 (0) | 4 (5) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3) | 4 (4) | 5 (5) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 13 (13) | 19 (19) | 18 (18) | 25 (26)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 5 (6) | 8 (9) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 10 (15) | 7 (11) | 19 (27) | 17 (35)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 0 (0) | 4 (4) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 3 (6) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (5) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Illness (General disorders) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Blood albumin decreased (Investigations) | 1 (2) | 2 (2) | 0 (0) | 3 (6) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 1 (4) | 2 (2) | 4 (9) | 2 (3)
Blood glucose increased (Investigations) | 2 (2) | 2 (4) | 0 (0) | 3 (4) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 3 (3) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0) | 3 (6) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 1 (1)
Lymphoedema (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT04177108/Prot_SAP_000.pdf